CLINICAL TRIAL: NCT03791086
Title: The BRIDGE Study - Bronchiectasis Research Involving Databases, Genomics and Endotyping. An EMBARC2 and EMBARC3 Study
Brief Title: The BRIDGE Study - Bronchiectasis Research Involving Databases, Genomics and Endotyping
Acronym: BRIDGE
Status: Recruiting | Type: Observational
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, James Chalmers, Professor, University of Dundee
Other Study IDs: 2017RC11
Record Dates: First submitted 2018-12-29; First posted 2019-01-02 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA Serum Sputum and sputum supernatant Urine Nasal swabs Nasal biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bronchiectasis: Adult patients with bronchiectasis meeting the inclusion criteria.

SUMMARY:
Bronchiectasis is a complex heterogeneous disorder. Treatment is challenging and many recent randomized controlled trials have been negative. It is believed that bronchiectasis as a broad diagnosis incorporates multiple different patient subgroups (also known as phenotypes) and molecular entities (referred to as endotypes). This study aims to phenotype and endotype bronchiectasis during stable disease and exacerbations, to develop strategies for personalised medicine.

Primary Objective To determine molecular endotypes of bronchiectasis which can guide response to treatment.

Secondary Objectives

1. To determine molecular endotypes of stable bronchiectasis
2. To determine the causes and inflammatory profiles of bronchiectasis exacerbations
3. To validate candidate biomarkers of stable and exacerbation endotypes to use in stratified medicine
4. To perform in-vivo or in-vitro proof of concept studies using phenotypic data to identify patient populations likely to benefit in future randomized controlled trials

This is an observational cohort study that will aim to identify patient subgroups and link these with meaningful clinical outcomes.

DETAILED DESCRIPTION:
Background: Bronchiectasis is a common disabling and heterogeneous disease that has been neglected in terms of basic and clinical research. Recent controlled trials have failed to achieve their primary end-points, likely because the optimal patient population to benefit from antibiotic, mucoactive and anti-inflammatory drugs has not been identified. This study aims to explore the clinical, microbiological, inflammatory and functional heterogeneity of the disease with the aim of identifying patient endotypes for stratified medicine.

Study aims and objectives

1. To determine the molecular endotypes of bronchiectasis during stable disease
2. To determine the causes and inflammatory profiles of bronchiectasis exacerbations
3. To validate candidate biomarkers of stable and exacerbation endotypes to use in stratified medicine
4. To perform in-vivo or in-vitro proof of concept studies using phenotypic data to identify patient populations likely to benefit in future randomized controlled trials Study Design: Observational Cohort study

Study methods:

Patients with bronchiectasis will be recruited into an observational study, the objectives of which will be to:

Aim 1 will define and validate endotypes of stable bronchiectasis by studying up to 1000 patients with bronchiectasis. Clinical data, sputum microbiome, sputum proteomics, and systemic and sputum inflammatory marker measurement will be incorporated for analysis. A sub-study (n=200) will be performed using air liquid interface culture of primary airway epithelial cells. Patients will have brushings of the inferior nasal turbinate with assessment of % ciliation, ciliary beat frequency and pattern by high speed video microscopy before and after culture.

Aim 2 will replicate the phenotyping approach to stable patients with 160 patients during exacerbation. This will identify changes from baseline in microbiota, proteomic and other markers associated with onset of exacerbation and allow classification of clusters of exacerbation.

Aim 3, we will externally validate candidate phenotype/endotypes in registered ethically approved external biobanks and aim to demonstrate that validated markers to be linked to potential treatment responses for use in stratified medicine trials.

In total we will recruit 1000 patients for study. These patients will attend the Clinical Research Centre at one of the participating study centres at least once and undergo sampling along with collecting of clinical data. Patients will be asked to consent for their samples to be linked to data held on the EMBARC registry.

Nature of outputs and outcomes/results expected:

This study will aim to establish detailed endotypes in bronchiectasis which can guide response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* A previous CT scan showing bronchiectasis along with compatible clinical syndrome of cough, sputum production and/or recurrent respiratory tract infections.
* A primary diagnosis of bronchiectasis made by a respiratory physician
* At the screening visit the individual will have been clinically stable for 4 weeks indicated by the lack of any treatment with antibiotics or corticosteroids for a pulmonary exacerbation in the previous 4 weeks.

Exclusion Criteria:

* Inability to give informed consent
* <18years of age
* Patients with active tuberculosis
* Treatment with antibiotics or corticosteroids for a pulmonary exacerbation in the previous 4 weeks
* Bronchiectasis due to cystic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of exacerbations | up to 3 years
  Worsening of respiratory symptoms as defined by the EMBARC/BRR definition- Eur Respir J. 2017 Jun 8;49(6). pii: 1700051.

SECONDARY OUTCOMES:
Time to first exacerbation | 3 years
  Time to first event after enrolment as defined by the EMBARC/BRR definition- Eur Respir J. 2017 Jun 8;49(6). pii: 1700051.
Quality of life- the quality of life bronchiectasis questionnaire (QOL-B) | 3 years
  Validated questionnaire
Quality of life- the St Georges Respiratory Questionnaire (SGRQ) | 3 years
  Validated questionnaire
Quality of life- The Bronchiectasis impact measure (BIM) | 3 years
  Questionnaire undergoing validation
Quality of life- The Bronchiectasis Health Questionnaire (BHQ) | 3 years
  Validated questionnaire
Forced expiratory volume in 1 second (FEV1) | 3 years
  Spirometry
Severity of disease (the bronchiectasis severity index) | 3 years
  Validated severity assessment tool
Hospitalisation for severe exacerbations | 3 years
  Admission to hospital for an exacerbation meeting the EMBARC/BRR exacerbation definition
All cause mortality | 3 years
  Survival during the study
Infection with Pseudomonas aeruginosa | 3 years
  Defined as isolation in sputum culture or bronchoalveolar lavage meeting the criteria for chronic infection- Ann Am Thorac Soc. 2015 Nov;12(11):1602-11.
Sputum volume | 3 years
  Measured in millilitres per day

CONTACTS AND LOCATIONS:
Overall Officials: James D Chalmers, MD, PhD, Principal Investigator — GSK/British Lung Foundation Chair of Respiratory Research
Locations (1):
- University of Dundee, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from EMBARC supported studies will be made available to researchers. Application for EMBARC data can be made on our website. Further information is available at www.bronchiectasis.eu/dataaccess
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Available following the study subject to approval by the scientific committee as detailed at www.bronchiectasis.eu/dataaccess
Access Criteria: Approval of an analysis protocol by an independent scientific committee

REFERENCES:
- [Derived] Choi H, Hughes C, Eke Z, Shuttleworth M, Shteinberg M, Polverino E, Goeminne PC, Welte T, Blasi F, Shoemark A, Long MB, Aliberti S, Haworth CS, Ringshausen FC, Loebinger MR, Lorent N, Chalmers JD. Clinical Efficacy of Serum Antiglycopeptidolipid Core IgA Antibody Test for Screening Nontuberculous Mycobacterial Pulmonary Disease in Bronchiectasis: A European Multicenter Cohort Study. Chest. 2025 May;167(5):1300-1310. doi: 10.1016/j.chest.2024.10.029. Epub 2024 Oct 28. PMID 39490969